CLINICAL TRIAL: NCT06475729
Title: A Bioequivalence Study of Subcutaneous Injections of Citrate-Free Mirikizumab Solution Using a 1-mL Autoinjector and an Investigational 2-mL Autoinjector in Healthy Participants
Brief Title: A Bioequivalence Study of Citrate Free Mirikizumab (LY3074828) in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18852; I6T-MC-AMCB (Other: Eli Lilly and Company)
Record Dates: First submitted 2024-06-21; First posted 2024-06-26 (Actual); Results first posted 2025-12-30 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Healthy
MeSH Terms: interventions — mirikizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 200 mg Mirikizumab (Test) (Experimental): Participants received 200 mg mirikizumab test formulation, 1 × 2-mL SC injections of 100 mg/mL citrate-free mirikizumab administered into arm/thigh/abdomen on day 1.
  Interventions: Drug: Citrate-Free Mirikizumab
- 200 mg Mirikizumab (Reference) (Experimental): Participants received 200 milligrams (mg) mirikizumab reference formulation, 2 × 1-milliliter (mL) subcutaneous (SC) injections of 100 mg/mL citrate-free mirikizumab administered into arm/thigh/abdomen on day 1.
  Interventions: Drug: Citrate-Free Mirikizumab

INTERVENTIONS:
Drug: Citrate-Free Mirikizumab — Administered SC
  Other Names: LY3074828

SUMMARY:
The purpose of this study is to evaluate the amount of mirikizumab (test) that gets into the blood stream and how long it takes the body to get rid of it, when given via autoinjector, an injection under the skin, compared to mirikizumab (reference) solution given via autoinjector.

Screening is required within 35 days prior to enrollment. For each participant, the total duration for of the clinical trial will be about 15 weeks, including screening.

ELIGIBILITY:
Inclusion Criteria:

Type of participant and disease characteristics

1. Overtly healthy males and females as determined by medical evaluation including:

   * Medical history,
   * Physical examination,
   * Clinical laboratory tests,
   * Electrocardiogram (ECG),
   * Vital signs

   Note: participants may have chronic, stable medical conditions that, in the investigator's opinion, will not place the participant at increased risk by participating in the study, and will not interfere with interpretation of the data.
2. Have clinical laboratory test results:

   * Within normal reference range for the population, or
   * Within normal reference range for the investigative site, or
   * Results with acceptable deviations that are judged to be not clinically significant by the investigator.

   Weight
3. Have a body mass index (BMI) within the range of 18.0 to 34.0 kilograms per milligram squared (km/m^2), inclusive.

   Exclusion Criteria:

   Participants are excluded from the study if any of the following criteria apply:

   Medical conditions
4. Have significant allergies to humanized monoclonal antibodies or known allergies to citrate-free mirikizumab, related compounds or any components of the formulation.
5. Have significant previous or current history of comorbidities capable of significantly altering the absorption, metabolism, or elimination of drugs; of constituting a risk when taking the investigational product; or of interfering with the interpretation of data.
6. Have clinically significant multiple or severe drug allergies, or intolerance to topical corticosteroids, or severe post-treatment hypersensitivity reactions.
7. Have a diagnosis or history of malignant disease within 5 years prior to baseline.

   Prior/concomitant therapy
8. Intend to use over-the-counter or prescription medication, including herbal medications and traditional medications, within 7 days prior to dosing.
9. Have received treatment with biologic agents, such as monoclonal antibodies, including marketed drugs, within 3 months or 5 half-lives, whichever is longer, prior to dosing.
10. Have ever received anti-interleukin (IL)-12p40 antibodies or anti-IL-23p19 antibodies, for any indication, including investigational use.
11. Have received any live vaccine (that is, live attenuated) within less than 4 weeks or inactivated vaccine within less than 2 weeks before randomization.

    Prior/concurrent clinical study experience
12. Are currently enrolled in a clinical study involving an investigational product or any other type of medical research judged not to be scientifically or medically compatible with this study.
13. Have participated in a clinical study involving an investigational product within the last 30 days or 5 half-lives, whichever is longer, prior to screening. If the clinical trial involved treatment with biologic agents, such as monoclonal antibodies, including marketed drugs, at least 3 months or 5 half-lives, whichever is longer, should have elapsed prior to dosing.
14. Have previously completed or withdrawn from this study or any other study investigating mirikizumab, and have previously received mirikizumab.

    Diagnostic assessments
15. Have a current infection with hepatitis C virus.
16. Have a current infection with hepatitis B virus.
17. Have a current or recent acute, active infection.
18. Have had any of the following types of infection within 3 months prior to screening or develops any of these infections before the randomization:

    1. Serious: Requiring hospitalization, or intravenous (IV) or equivalent oral antibiotic treatment, or both.
    2. Opportunistic: As defined in Winthrop et al. 2015. Note: Herpes zoster is considered active and ongoing until all vesicles are dry and crusted over.
    3. Chronic: Duration of symptoms, signs, and/or treatment of 6 weeks or longer.
    4. Recurring: Including, but not limited to, herpes simplex, herpes zoster, recurring cellulitis, chronic osteomyelitis.
19. Show evidence of active or latent tuberculosis (TB).

    Other exclusion criteria
20. Have alcohol intake that exceeds recommended average weekly alcohol consumption limits per local regulation, or an amount deemed significant by the investigator.
21. Smoke more than 10 cigarettes per day, or equivalent, or are unable to abide by investigative site smoking restrictions.
22. In the opinion of the investigator or sponsor, are unsuitable for inclusion in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 498 (Actual)
Dates: Start 2024-06-24 (Actual); Primary Completion 2024-12-27 (Actual); Study Completion 2024-12-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 : Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (6):
- United States (6):
  - CenExel ACT, Anaheim, California
  - Fortrea Clinical Research Unit, Daytona Beach, Florida
  - Clinical Pharmacology of Miami, Miami, Florida
  - QPS Missouri, Springfield, Missouri
  - Fortrea Clinical Research Unit, Dallas, Texas
  - Fortrea Clinical Research Unit, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Otani Y, Payne CD, Loftus EV Jr, D'Haens G, Ben Horin S, Upadhya K A, Todd K, Pellanda P, Shi G, Zhang X. One Subcutaneous 2-ml Injection of Mirikizumab is Bioequivalent to Two 1-ml Subcutaneous Injections in Healthy Participants. Adv Ther. 2025 Nov 28. doi: 10.1007/s12325-025-03422-1. Online ahead of print. PMID 41313544

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 200 mg Mirikizumab (Reference) | 200 mg Mirikizumab (Test)
Started | 249 | 249
All Participants Who Were Exposed to Study Intervention (Safety Population) | 240 | 244
Completed | 237 | 241
Not Completed | 12 | 8
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Randomized but did not receive any dose | 3 | 2
Not completed — Lost to Follow-up | 1 | 2
Not completed — Physician Decision | 5 | 2
Not completed — Adverse Event | 1 | 1

BASELINE CHARACTERISTICS:
Population: All participants who were exposed to study intervention (Safety Population).
Groups:
- 200 mg Mirikizumab (Reference): Participants received 200 mg mirikizumab reference formulation, 2 × 1-mL SC injections of 100 mg/mL citrate-free mirikizumab administered into arm/thigh/abdomen on day 1.
- Total: Total of all reporting groups
Arm/Group | 200 mg Mirikizumab (Reference) | 200 mg Mirikizumab (Test) | Total
Number analyzed (Participants) | 240 | 244 | 484
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.7 (11.6) | 42.4 (12.5) | 42.5 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 112 | 135 | 247
  Male | 128 | 109 | 237
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 111 | 108 | 219
  Not Hispanic or Latino | 129 | 136 | 265
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 8 | 10 | 18
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 52 | 56 | 108
  White | 177 | 174 | 351
  More than one race | 3 | 2 | 5
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 240 | 244 | 484

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics (PK): Maximum Observed Drug Concentration (Cmax) of Mirikizumab
Description: Cmax of Mirikizumab is reported.
Time Frame: Day 1: Predose, 72, 120, 192, 264, 360, 528, 696, 1032, 1368, 1704 hours post-dose.
Population: All enrolled participants who received a full dose of study intervention and have evaluable PK data for this outcome according to the study intervention actually received.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram per milliliter (ug/mL)
Arm/Group | 200 mg Mirikizumab (Reference) | 200 mg Mirikizumab (Test)
Number analyzed (Participants) | 238 | 243
microgram per milliliter (ug/mL) | 12.9 (40) | 13.5 (39)
Statistical Analysis 1: Comparison: 200 mg Mirikizumab (Reference) vs 200 mg Mirikizumab (Test); Test type: Equivalence — Log-transformed PK parameters were analyzed using a fixed-effects model. Bioequivalence will be concluded if the 2-sided 90% Confidence Interval is completely contained within the interval (0.80, 1.25); Ratio of Geometric least squares mean = 1.039, 90% CI 2-sided [0.9853 to 1.0956]

2. Primary Outcome: PK: Area Under the Concentration Versus Time Curve From Time Zero to Infinity (AUC [0-∞]) of Mirikizumab
Description: AUC [0-∞] of Mirikizumab is reported.
Time Frame: Day 1: Predose, 72, 120, 192, 264, 360, 528, 696, 1032, 1368, 1704 hours post-dose.
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram*day per milliliter (ug*day/mL)
Arm/Group | 200 mg Mirikizumab (Reference) | 200 mg Mirikizumab (Test)
Number analyzed (Participants) | 238 | 243
microgram*day per milliliter (ug*day/mL) | 225 (41) | 228 (41)
Statistical Analysis 1: Comparison: 200 mg Mirikizumab (Reference) vs 200 mg Mirikizumab (Test); Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of Geometric least squares mean = 1.011, 90% CI 2-sided [0.9564 to 1.0685]

3. Primary Outcome: PK: Area Under the Concentration Versus Time Curve From Time 0 to the Last Measurable Concentration (AUC [0-tlast]) of Mirikizumab
Description: AUC [0 to tlast] of Mirikizumab is reported.
Time Frame: Day 1: Predose, 72, 120, 192, 264, 360, 528, 696, 1032, 1368, 1704 hours post-dose.
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram*day per milliliter (ug*day/mL)
Arm/Group | 200 mg Mirikizumab (Reference) | 200 mg Mirikizumab (Test)
Number analyzed (Participants) | 238 | 241
microgram*day per milliliter (ug*day/mL) | 220 (40) | 223 (41)
Statistical Analysis 1: Comparison: 200 mg Mirikizumab (Reference) vs 200 mg Mirikizumab (Test); Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of Geometric least squares mean = 1.011, 90% CI 2-sided [0.9568 to 1.0678]

ADVERSE EVENTS:
Time Frame: Baseline up to Day 74
Description: All participants who were exposed to study intervention (Safety Population). Participants were analyzed according to the intervention they actually received.
Arm/Group | 200 mg Mirikizumab (Reference) | 200 mg Mirikizumab (Test)
All-Cause Mortality (participants affected / at risk) | 0/240 | 0/244
Serious Adverse Events (participants affected / at risk) | 0/240 | 0/244
Other Adverse Events (participants affected / at risk) | 55/240 | 48/244
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 200 mg Mirikizumab (Reference) (N=240) | 200 mg Mirikizumab (Test) (N=244)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (2)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 2 (2)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (4) | 2 (2)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1)
Chills (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 1 (1)
Injection site bruising (General disorders) | 2 (3) | 1 (1)
Injection site pain (General disorders) | 1 (1) | 0 (0)
Injection site reaction (General disorders) | 4 (6) | 5 (5)
Pain (General disorders) | 1 (1) | 1 (1)
Peripheral swelling (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Vessel puncture site bruise (General disorders) | 2 (2) | 1 (1)
Hepatitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Covid-19 (Infections and infestations) | 0 (0) | 2 (2)
Escherichia urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Furuncle (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 1 (1)
Pharyngitis (Infections and infestations) | 3 (3) | 2 (2)
Pharyngitis streptococcal (Infections and infestations) | 1 (1) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 2 (2)
Tooth infection (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 4 (4) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Clavicle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pulmonary contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 1 (1)
Blood potassium increased (Investigations) | 1 (1) | 1 (1)
Sars-cov-2 test positive (Investigations) | 0 (0) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 3 (4) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Dizziness (Nervous system disorders) | 2 (2) | 1 (1)
Headache (Nervous system disorders) | 9 (9) | 12 (14)
Loss of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 2 (2) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Abnormal dreams (Psychiatric disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 2 (2) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2024-09-24): https://cdn.clinicaltrials.gov/large-docs/29/NCT06475729/Prot_000.pdf
  • Statistical Analysis Plan (2024-06-06): https://cdn.clinicaltrials.gov/large-docs/29/NCT06475729/SAP_001.pdf